CLINICAL TRIAL: NCT02454530
Title: PROPHYLACTIC TREATMENT FOR CHEMO-INDUCED NEUTROPENIA. USE OF G-CSF BIOSIMILAR (NIVESTIM(REGISTERED)) ACCORDING TO THE CHEMOTHERAPY CONTEXT: ADJUVANT VERSUS METASTATIC.
Brief Title: Use of Biosimilar Nivestim® to Prevent Chemo-induced Neutropenia. Real Life Study
Acronym: VISTA
Status: Terminated | Type: Observational
Why Stopped: The study was stopped due to the judicial liquidation of the CRO in charge of this study.
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: VISTA; C1121007 (Other: Alias Study Number)
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-03

CONDITIONS: Chemotherapy-Induced Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients treated with Nivestim®
  Interventions: Biological: Nivestim®

INTERVENTIONS:
Biological: Nivestim®

SUMMARY:
The aim of this study is to describe in real-life conditions the determinants of use of GCSF (Granulocyte Colony-Stimulating Factor) Nivestim® in primary or secondary prophylaxis and in patients receiving chemotherapy for solid tumour according to the chemotherapy context: adjuvant or metastatic setting.

DETAILED DESCRIPTION:
This is a longitudinal, observational, prospective, multicentre, cohort study, conducted in France among a representative sample of public and/or private hospital-based oncologists.

Data will be collected by the investigator during three visits using data available in the patient medical record and obtained from patient questioning and clinical examination performed during the consultations:

* Baseline visit: prescription of Nivestim®.
* Follow-up visit: during the first cycle of chemotherapy after the first course of Nivestim®.
* Final visit: after the last cycle of chemotherapy or 16-18 weeks after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years, seen by the oncologist for chemotherapy for solid tumour.
* Patients for whom the oncologist has decided the initiation of G-CSF biosimilar treatment (Nivestim®) in primary or secondary prophylaxis.
* Patients informed about the computer processing of their medical data and their right of access and correction.

Exclusion Criteria:

* Patients with contraindication of use of Nivestim®.
* Patients with haematological malignancy including Myelodysplasia and Chronic myeloid leukemia treated or untreated.
* Patients participating or having participated in the previous month in a clinical trial.
* Patients refusing to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumour treated with cytotoxic chemotherapy and for whom a prophylactic treatment with G-CSF biosimilar (Nivestim®) is initiated
Sampling Method: Non-Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (90):
- France (90):
  - Clinique Rambot La Provençale Tour d'Aygosi, Aix-en-Provence
  - Centre Hospitalier du Pays d'Aix Service d'Hématologie - Oncologie, Aix-en-Provence
  - ICO Centre Paul Papin Service d'Oncologie Médicale, Angers
  - CHU - Hôtel-Dieu Service Hépato-Gastro-entérologie, Angers
  - CH d'Armentières Service Oncologie, Armentières
  - Centre Marie Curie A l'attention de Laëtitia, Arras
  - Centre Hospitalier Service Oncologie, Auxerre
  - Clinique du Dr Maymard Service d'Oncologie, Bastia
  - Hôpital de Falconaja Furiani Service d'Oncologie, Bastia
  - Centre Hospitalier Philippe le Bon Service de Medecine Interne - 3e Etage, Beaune
  - CHU - Hôpital Jean Minjoz Service Oncologie Médicale, Besançon
  - Centre Hospitalier Service Onco-Hématologie, Béziers
  - Hôpital Avicenne Service Gastro-Entérologie, Bobigny
  - Clinique Tivoli, Bordeaux
  - Centre Hospitalier Service d'Oncologie, Boulogne-sur-Mer
  - CH de Fleyriat Service de Pneumologie, Bourg-en-Bresse
  - CH de Fleyriat Service Onco-Hématologie, Bourg-en-Bresse
  - Clinique Pasteur Lanroze Service Oncologie, Brest
  - Hôpital Augustin Morvan Institut de Cancérologie et d'Hématologie, Brest
  - Hôpital Morvan - CHU Institut de Cancérologie et d'Hématologie, Brest
  - Hôpital Louis Pradel Service Pneumologie - Centre des Maladies Orphelines, Bron
  - Centre François Baclesse Oncologie Médicale. Pathologie Mammaire et Recherche Clinique, Caen
  - Centre Hospitalier Service d'Oncologie, Carcassonne
  - Centre Hospitalier de Carcassonne Service d'Oncologie, Carcassonne
  - Medipole de Savoie Service Oncologie, Challes-les-Eaux
  - Médipole de Savoie, Challes-les-Eaux
  - CH William Morey Service d'Oncologie Médicale, Chalon-sur-Saône
  - CHP du Cotentin - Site de Cherbourg Service d'Oncologie, Cherbourg
  - Centre Hospitalier de Cholet Service d' Oncologie Médicale, Cholet
  - Centre Hospitalier de Cholet Service d'Hepato-Gastro-Enterologie, Cholet
  - Centre hospitalier Louis Pasteur Service de Pneumologie, Colmar
  - Hôpital Louis Pasteur Service de Pneumologie - Médecine F, Colmar
  - Centre de Radiothérapie GIE CROM, Compiègne
  - CHU de Dijon - Hôpital du Bocage Service Hépato-Gastro-Entérologie, Dijon
  - Centre Hospitalier de la Dracénie Service d'Oncologie, Draguignan
  - Centre Hospitalier Emile Durkheim Service Oncologie, Épinal
  - Clinique Chirurgicale Pasteur Service Oncologie Médicale, Évreux
  - CHI Fréjus Saint Raphaël Service d'Oncologie Médicale, Fréjus
  - CHI des Alpes du sud Site de Gap Muret Hôpital de Jour - Oncologie, Gap
  - Centre Hospitalier Service d'Oncologie, Gonesse
  - Centre Hospitalier Service Onco-Hématologie, Le Mans
  - Centre de Radiothérapie Hartmann, Levallois-Perret
  - Institut Franco Britannique Service Oncologie Médicale, Levallois-Perret
  - Clinique Hartman Service de Radiothérapie, Levallois-Perret
  - Clinique Hartmann Service Oncologie, Levallois-Perret
  - CHRU Lille - Hôpital Huriez Unité d'Oncologie Médicale, Lille
  - CHU Dupuytren Limoges Service d'Oncologie, Limoges
  - Centre Hospitalier Service de Médecine 2 - Hôpital de jour, Lons-le-Saunier
  - Centre Léon Bérard Service d'Oncologie Médicale, Lyon
  - Hôpital Privé Jean Mermoz Service d'Oncologie Médicale, Lyon
  - CH Saint-Joseph et Saint-Luc Service de Gastro-Entérologie, Lyon Cedez 07
  - Centre Hospitalier Privé Clairval Service de Cancérologie, Marseille
  - Hôpital Nord Service d'Oncologie Multidisciplinaires et Innovations Thérapeutiques, Marseille
  - Clinique Claude Bernard Service de Chimiothérapie, Metz
  - Clinique Claude Bernard Service Chimiothérapie, Metz
  - Centre Hospitalier Layne Service d'Oncologie, Mont-de-Marsan
  - Centre Hospitalier de Belfort-Montbéliard Site du Mittan-Oncologie et radiothérapie, Montbéliard
  - Clinique Clementville Service d'Oncologie, Montpellier
  - CHU Montpellier - Hôpital Arnaud de Villeneuve Service de Cancérologie, Montpellier
  - Centre Hospitalier Emile Muller, Mulhouse
  - CH de Mulhouse - Hôpital Emile Muller Hôpital de Jour - Oncologie, Mulhouse
  - Polyclinique de Gentilly Service Oncologie Médicale, Nancy
  - CHU - Hôpital Hôtel Dieu Unité de Gastroentérologie, Nantes
  - CHU de Nantes - Hôpital Laënnec Service d'Oncologie Médicale, Nantes
  - Centre Hospitalier de Narbonne Oncologie / Hématologie, Narbonne
  - Hôpital Américain, Neuilly-sur-Seine
  - Institut Mutualiste Montsouris Service Oncologie Médicale, Paris
  - Clinique Alleray Labrouste Service d'Oncologie Médicale, Paris
  - Hôpital Européen Georges Pompidou Service d'Oncologie Médicale, Paris
  - Hôpital Européen Georges Pompidou Service Oncologie Médicale - 4e étage (ascenseur B), Paris
  - Hôpital Bichat Claude Bernard Service Hépato-Gastroentérologie et Cancérologie Digestive, Paris
  - Hôpital Tenon Service d'oncologie médicale, Paris
  - Centre Hospitalier Service d'Oncologie, Perpignan
  - Centre Hospitalier Service de Pneumologie, Perpignan
  - Centre Hospitalier Annecy Genevois Service Pneumologie, Pringy
  - Centre Hospitalier de la region d'Annecy Pole Medecine, Pringy
  - CH de Cornouaille Service d'Oncologie Médicale, Quimper
  - Institut Jean Godinot, Reims
  - Clinique de l'Europe Unité d'Oncologie, Rouen
  - Hôpital de Saint-Avold Service Oncologie II, Saint-Avold
  - Clinique François 1er, Saint-Dizier
  - Centre Hospitalier Privé Saint Grégoire Service d'Oncologie - Radiothérapie, Saint-Grégoire
  - Centre Hospitalier Privé Saint-Grégoire Service d'Oncologie - Radiothérapie, Saint-Grégoire
  - Centre Clinical Service d'Oncologie-Radiothérapie, Soyaux
  - Centre de Radiothérapie SCP Strasbourg Oncologie Libérale, Strasbourg
  - Hôpital Bel Air Service Pneumologie, Thionville
  - Hôpital de Thionville Service Oncologie Médicale, Thionville
  - Hôpital Rangueil Service d'Oncologie Médicale Digestive et Gynécologique, Toulouse
  - Clinique Pasteur, Toulouse
  - Hôpital Bretonneau Service d'Oncologie Médicale, Tours

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2014 and September 2016, 102 public and/or private hospital-based oncologists included 1160 patients with solid tumor treated with cytotoxic chemotherapy and for whom a prophylactic treatment with G-CSF (Granulocyte Colony-Stimulating Factor) biosimilar (Nivestim®) was initiated. The study was conducted in France.
Groups:
- Adjuvant Chemotherapy: Participants who were receiving chemotherapy for solid tumor in the adjuvant setting and for whom a prophylactic treatment with G-CSF (Granulocyte Colony-Stimulating Factor) biosimilar (Nivestim®) was initiated (maximum duration was 15 days) were observed for a maximum of 2.25 years in this study.
- Metastatic Chemotherapy: Participants who were receiving chemotherapy for solid tumor in the metastatic setting and for whom a prophylactic treatment with G-CSF biosimilar (Nivestim®) was initiated (maximum duration was 10 days) were observed for a maximum of 2.25 years in this study.
Period: Overall Study
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Started | 552 | 608
Completed | 482 | 481
Not Completed | 70 | 127
Not completed — Other | 8 | 13
Not completed — Missing information | 56 | 69
Not completed — Death | 2 | 41
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who received at least one dose of Nivestim® and did not had a major deviation from the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy | Total
Number analyzed (Participants) | 551 | 603 | 1154
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Here, 'Number analyzed' signifies number of participants evaluable for this baseline characteristics.
  years
    number analyzed (Participants) | 551 | 599 | 1150
    (all) | 60.3 (12.1) | 65.0 (11.0) | 62.7 (11.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 399 | 324 | 723
  Male | 149 | 277 | 426
  Missing | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Level of Importance of Factors Determining the Use of Nivestim
Description: The factors which determined the use of Nivestim among participants included participant's sex, young participant, elderly participant, past history of infection, comorbidities, life expectancy, past history of febrile neutropenia and severe neutropenia, occupational activity, family activity and other important criteria. Percentage of participants were categorized based upon the level of importance under different categories which included very important, important, relatively important, not important and not applicable.
Time Frame: Inclusion visit (Week 1)
Population: Analysis population included all participants who received at least one dose of Nivestim and did not had a major deviation from the protocol. Here 'Number analyzed' signifies number of participants evaluable for specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 551 | 603
Percentage of participants
  Participant sex: Very important (VI): number analyzed (Participants) | 547 | 595
  Participant sex: Very important (VI) | 2.7 | 1.7
  Participant sex: Important: number analyzed (Participants) | 547 | 595
  Participant sex: Important | 11.2 | 7.2
  Participant sex: Relatively unimportant (RU): number analyzed (Participants) | 547 | 595
  Participant sex: Relatively unimportant (RU) | 24.5 | 22.5
  Participant sex: Not important (NI): number analyzed (Participants) | 547 | 595
  Participant sex: Not important (NI) | 52.3 | 58.2
  Participant sex: Not applicable (NA): number analyzed (Participants) | 547 | 595
  Participant sex: Not applicable (NA) | 9.3 | 10.4
  Young participant: VI: number analyzed (Participants) | 547 | 594
  Young participant: VI | 4.6 | 2.7
  Young participant: Important: number analyzed (Participants) | 547 | 594
  Young participant: Important | 17.2 | 9.3
  Young participant: RU: number analyzed (Participants) | 547 | 594
  Young participant: RU | 26.5 | 26.8
  Young participant: NI: number analyzed (Participants) | 547 | 594
  Young participant: NI | 24.5 | 27.1
  Young participant: NA: number analyzed (Participants) | 547 | 594
  Young participant: NA | 27.2 | 34.2
  Elderly participant: VI: number analyzed (Participants) | 543 | 596
  Elderly participant: VI | 22.3 | 20.8
  Elderly participant: Important: number analyzed (Participants) | 543 | 596
  Elderly participant: Important | 30.6 | 33.9
  Elderly Participant: RU: number analyzed (Participants) | 543 | 596
  Elderly Participant: RU | 12.9 | 13.3
  Elderly participant: NI: number analyzed (Participants) | 543 | 596
  Elderly participant: NI | 12.7 | 14.4
  Elderly participant: NA: number analyzed (Participants) | 543 | 596
  Elderly participant: NA | 21.5 | 17.6
  Past history of infection: VI: number analyzed (Participants) | 546 | 595
  Past history of infection: VI | 16.7 | 15.6
  Past history of infection: Important: number analyzed (Participants) | 546 | 595
  Past history of infection: Important | 22.5 | 25.7
  Past history of infection: RU: number analyzed (Participants) | 546 | 595
  Past history of infection: RU | 11.2 | 13.8
  Past history of infection: NI: number analyzed (Participants) | 546 | 595
  Past history of infection: NI | 17.2 | 17.6
  Past history of infection: NA: number analyzed (Participants) | 546 | 595
  Past history of infection: NA | 32.4 | 27.2
  Comorbidities: VI: number analyzed (Participants) | 546 | 594
  Comorbidities: VI | 19.6 | 20.4
  Comorbidities: Important: number analyzed (Participants) | 546 | 594
  Comorbidities: Important | 27.8 | 32.8
  Comorbidities: RU: number analyzed (Participants) | 546 | 594
  Comorbidities: RU | 15.6 | 15.0
  Comorbidities: NI: number analyzed (Participants) | 546 | 594
  Comorbidities: NI | 15.4 | 15.7
  Comorbidities: NA: number analyzed (Participants) | 546 | 594
  Comorbidities: NA | 21.6 | 16.2
  Life expectancy: VI: number analyzed (Participants) | 545 | 593
  Life expectancy: VI | 23.1 | 15.5
  Life expectancy: Important: number analyzed (Participants) | 545 | 593
  Life expectancy: Important | 26.4 | 31.4
  Life expectancy: RU: number analyzed (Participants) | 545 | 593
  Life expectancy: RU | 18.5 | 24.8
  Life expectancy: NI: number analyzed (Participants) | 545 | 593
  Life expectancy: NI | 14.5 | 15.2
  Life expectancy: NA: number analyzed (Participants) | 545 | 593
  Life expectancy: NA | 17.4 | 13.2
  Past history febrile neutropenia (FN): VI: number analyzed (Participants) | 546 | 596
  Past history febrile neutropenia (FN): VI | 29.9 | 29.7
  Past history FN: Important: number analyzed (Participants) | 546 | 596
  Past history FN: Important | 7.5 | 12.2
  Past history FN: RU: number analyzed (Participants) | 546 | 596
  Past history FN: RU | 7.1 | 7.0
  Past history FN: NI: number analyzed (Participants) | 546 | 596
  Past history FN: NI | 13.9 | 13.8
  Past history FN: NA: number analyzed (Participants) | 546 | 596
  Past history FN: NA | 41.6 | 37.2
  Past history of severe neutropenia (SN): VI: number analyzed (Participants) | 547 | 594
  Past history of severe neutropenia (SN): VI | 26.9 | 29.3
  Past history of SN: Important: number analyzed (Participants) | 547 | 594
  Past history of SN: Important | 16.1 | 19.2
  Past history of SN: RU: number analyzed (Participants) | 547 | 594
  Past history of SN: RU | 8.2 | 8.9
  Past history of SN: NI: number analyzed (Participants) | 547 | 594
  Past history of SN: NI | 11.9 | 10.9
  Past history of SN: NA: number analyzed (Participants) | 547 | 594
  Past history of SN: NA | 36.9 | 31.6
  Occupational activity: VI: number analyzed (Participants) | 546 | 595
  Occupational activity: VI | 2.6 | 1.8
  Occupational activity: Important: number analyzed (Participants) | 546 | 595
  Occupational activity: Important | 8.4 | 7.9
  Occupational activity: RU: number analyzed (Participants) | 546 | 595
  Occupational activity: RU | 28.0 | 22.4
  Occupational activity:NI: number analyzed (Participants) | 546 | 595
  Occupational activity:NI | 26.6 | 29.4
  Occupational activity: NA: number analyzed (Participants) | 546 | 595
  Occupational activity: NA | 34.4 | 38.5
  Family activity: VI: number analyzed (Participants) | 545 | 593
  Family activity: VI | 2.9 | 1.0
  Family activity: Important: number analyzed (Participants) | 545 | 593
  Family activity: Important | 15.2 | 13.0
  Family activity: RU: number analyzed (Participants) | 545 | 593
  Family activity: RU | 22.4 | 18.5
  Family activity: NI: number analyzed (Participants) | 545 | 593
  Family activity: NI | 26.4 | 28.8
  Family activity: NA: number analyzed (Participants) | 545 | 593
  Family activity: NA | 33.0 | 38.6
  Other VI/ Important criteria: number analyzed (Participants) | 95 | 129
  Other VI/ Important criteria | 17.2 | 21.4

2. Secondary Outcome: Number of Participants Who Continued Chemotherapy
Description: Chemotherapy is a type of cancer treatment that uses one or more anti-cancer drugs as a part of a standardize treatment regimen. Chemotherapy may be given with curative intent, or it may aim to prolong life or to reduce symptoms.
Time Frame: Follow-up visit (Week 3); End of study visit ( up to Week 19)
Population: Analysis population included all participants who received at least one dose of Nivestim and did not had a major deviation from the protocol. Here, 'Number analyzed' signifies number of participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 551 | 603
Participants
  Follow up visit: number analyzed (Participants) | 536 | 566
  Follow up visit | 514 | 524
  End of study visit: number analyzed (Participants) | 493 | 520
  End of study visit | 111 | 202

3. Secondary Outcome: Number of Participants Who Discontinued Chemotherapy
Time Frame: Follow-up visit (Week 3); End of study visit ( up to Week 19)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 551 | 603
Participants
  Follow up visit: number analyzed (Participants) | 536 | 566
  Follow up visit | 22 | 42
  End of study visit: number analyzed (Participants) | 493 | 520
  End of study visit | 482 | 502

4. Secondary Outcome: Number of Participants With Unplanned Discontinuation of Chemotherapy at Follow Up Visit
Time Frame: Follow-up visit (Week 3)
Population: Analysis population included all participants who received at least one dose of Nivestim and did not had a major deviation from the protocol. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for the specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 22 | 42
Participants | 10 | 36

5. Secondary Outcome: Number of Participants With Dose Reduction in Chemotherapy Due to Neutropenia
Description: Neutropenia is an abnormally low level of neutrophils (count of less than 1,500 neutrophils per microliter (microL) in blood) and was classified as Grade 1 (mild) with an absolute neutrophil count (ANC) of 1000-1500 cells per microL, Grade 2 (moderate) with an ANC of 500-1000 cells per microL, or Grade 3 (severe) with an ANC lower than 500 cells per microL.
Time Frame: Follow-up visit (Week 3)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 12 | 15
Participants | 0 | 1

6. Secondary Outcome: Number of Participants With Delayed Administration of Chemotherapy Cycle Due to Neutropenia
Description: as for outcome 5
Time Frame: Follow-up visit (Week 3)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 12 | 15
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Unplanned Discontinuation of Chemotherapy at the End of Study Visit
Description: The reasons for unplanned discontinuation of chemotherapy included neutropenia, febrile neutropenia, other toxicity, development of resistance to treatment and other. Also, one participant could have more than one reason for unplanned discontinuation.
Time Frame: End of study visit (up to Week 19)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 482 | 502
Participants | 39 | 136

8. Secondary Outcome: Number of Participants With Change in Chemotherapy Protocol at End of Study Visit
Description: Number of participants with change in chemotherapy protocol due to each conditions (neutropenia, febrile neutropenia, neutropenia/febrile neutropenia, other toxicity, neutropenia/other toxicity) has been reported in this outcome measure.
Time Frame: End of study visit (up to Week 19)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 86 | 118
Participants
  Neutropenia | 21 | 21
  Febrile neutropenia | 2 | 2
  Other toxicity | 57 | 89
  Neutropenia/Febrile neutropenia | 2 | 0
  Neutropenia/Other toxicity | 2 | 6
  Febrile neutropenia/Other toxicity | 2 | 0

9. Secondary Outcome: Number of Participants With Neutropenia and Febrile Neutropenia
Description: Neutropenia is an abnormally low level of neutrophils (count of less than 1,500 neutrophils per microL in blood) and was classified as Grade 1 (mild) with an ANC of 1000-1500 cells per microL, Grade 2 (moderate) with an ANC of 500-1000 cells per microL, or Grade 3 (severe) with an ANC lower than 500 cells per microL. The incidence of neutropenia (between follow up and final visit) were described from the questionnaire completed by the investigator during the final visit. Febrile neutropenia was defined as tympanic or axillary body temperature greater than (>) 38.5 degree celsius for >1 hour and ANC less than (<) 1.0 *10^9 neutrophils per liter. The incidence of febrile neutropenia were described from the questionnaire completed by the investigator during the follow-up and final visits. Only those categories which had atleast 1 abnormality have been reported in this outcome measure.
Time Frame: Follow-up visit (Week 3); End of study visit (up to Week 19)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 551 | 603
Participants
  Follow up visit: Febrile Neutropenia: number analyzed (Participants) | 535 | 565
  Follow up visit: Febrile Neutropenia | 21 | 19
  Follow up visit: Neutropenia: number analyzed (Participants) | 535 | 565
  Follow up visit: Neutropenia | 21 | 21
  Final visit: Febrile Neutropenia: number analyzed (Participants) | 491 | 515
  Final visit: Febrile Neutropenia | 9 | 16
  Final visit: Neutropenia: number analyzed (Participants) | 491 | 515
  Final visit: Neutropenia | 63 | 75

10. Secondary Outcome: Change From Inclusion Visit in Disease Status as Measured by Number of Neutrophil Cells (Neutrophils), Platelet Count and Leukocyte Count at End of Study
Description: Change in the disease status of the participant was measured by the change in the count of neutrophils (NPs), platelets and leukocytes as reported in this outcome measure.
Time Frame: Inclusion visit (Week 1), End of study visit (up to Week 19)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 551 | 603
gram per liter (g/L)
  NP count at Inclusion Visit: number analyzed (Participants) | 522 | 592
  NP count at Inclusion Visit | 4.6 (15.4) | 5.3 (16.9)
  Change in NP count: number analyzed (Participants) | 451 | 488
  Change in NP count | -0.2 (10.9) | 1.8 (33.2)
  Platelet count at Inclusion Visit: number analyzed (Participants) | 528 | 594
  Platelet count at Inclusion Visit | 279.7 (103.6) | 261.4 (122.9)
  Change in platelet count: number analyzed (Participants) | 456 | 491
  Change in platelet count | -31.9 (117.0) | -43.4 (127.2)
  Leukocyte count at Inclusion Visit: number analyzed (Participants) | 523 | 594
  Leukocyte count at Inclusion Visit | 7.6 (26.4) | 6.7 (9.4)
  Change in leukocyte count: number analyzed (Participants) | 451 | 489
  Change in leukocyte count | -0.1 (13.3) | 1.5 (17.7)

11. Secondary Outcome: Change From Inclusion Visit in Disease Status as Measured by Participants Performance Status at End of Study
Description: The Karnofsky performance scale was used for rating participant activities of daily living. The KPS scores range from 0 to 100. A higher score means the participant is better able to carry out daily activities. The lower the Karnofsky score, the worse the survival for most serious illnesses. The score ranges included as 100 (Normal; no complaints), 90 (Able to carry on normal activity), 80 (Normal activity with effort), 70 (Cares for self; unable to carry on normal activity), 60 (Requires occasional assistance, but is able to care), 50 (Requires considerable assistance and frequent medical care), 40 (Disabled; requires special care), 30 (Severely disabled), 20 (Very sick; hospital admission necessary), 10 (Moribund; fatal processes progressing rapidly) and 0 (Dead).
Time Frame: Inclusion visit (Week 1); End of study visit (up to Week 19)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 315 | 318
score on a scale | -2.7 (11.0) | -9.1 (20.7)

12. Secondary Outcome: Change From Inclusion Visit in Disease Status as Measured by Haemoglobin Level at End of Study Visit
Description: Change in the disease status of the participant was measured by the change in the hemoglobin level as reported in this outcome measure.
Time Frame: Inclusion visit (Week 1), End of study visit (up to Week 19)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dl)
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 457 | 493
grams per deciliter (g/dl) | -1.2 (1.6) | -0.9 (1.7)

13. Secondary Outcome: Pain Experienced by Participant During Injection of Nivestim as Assessed by Pain at the Injection Site
Description: Pain experienced by participant at the injection site was measured on a scale 0 to 10 (0 = no pain to 10 = maximum pain), where higher score indicates maximum pain.
Time Frame: End of study visit (up to Week 19)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 458 | 469
unit on a scale | 2.0 (2.0) | 2.0 (2.0)

14. Secondary Outcome: Number of Participants With Chemotherapy Satisfaction as Per Doctor Assessment After Chemotherapy Treatment
Description: Participant's satisfaction after the chemotherapy treatment was assessed by the doctor and was categorized under the 4 categories as very satisfied, satisfied, not very satisfied and dissatisfied.
Time Frame: End of study visit (up to Week 19)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 472 | 478
Participants
  Very satisfied | 158 | 113
  Satisfied | 276 | 330
  Not very satisfied | 25 | 30
  Dissatisfied | 13 | 5

15. Secondary Outcome: Number of Participants Who Wished to Again Have Nivestim Treatment If Necessary
Time Frame: End of study visit (up to Week 19)
Population: Analysis population included all participants who received at least one dose of Nivestim and did not have a major deviation from the protocol. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for the specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 460 | 467
Participants | 424 | 428

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in participants who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment Emergent Adverse Event (TEAE) was adverse event that started or worsened in severity after Inclusion visit up to end of study visit (up to Week 19). AEs included both serious and non-serious adverse event. If a participant who reported an SAE also reported an AE that was not serious, that would count as 1 participant in the total number of participants reporting AEs.
Time Frame: Inclusion visit (Week 1) up to end of study visit (up to Week 19)
Population: The safety population included all participants who received at least one dose of Nivestim during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
Number analyzed (Participants) | 552 | 608
Participants
  AEs | 80 | 68
  SAEs | 3 | 2

17. Other Pre Specified Outcome: Number of Participants in Different Profiles Receiving Treatment With Nivestim
Description: Classification of participants into three different profiles were established by level of importance of the determining factors for the use of Nivestim and was categorized as profile 1= not applicable, profile 2= relatively unimportant and profile 3 = not important. A multiple correspondence analysis was conducted on the whole analysis population in order to identify possible different patient profiles. None of these profiles could have been associated to a type of chemotherapy (adjuvant or metastatic).
Time Frame: End of study visit (up to Week 19)
Population: Analysis population included all participants who received at least one dose of Nivestim and did not had a major deviation from the protocol and who did not had any missing importance level for the determining factors for the use of Nivestim. Here, "Overall Number of Participants Analyzed"=number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Adjuvant or Metastatic Chemotherapy: Participants with previous solid tumour who were prescribed Nivestim at the inclusion visit (Week 1), and were receiving adjuvant or metastatic type of chemotherapy after first course of Nivestim (maximum duration was 15 days for adjuvant chemotherapy and 10 days for metastatic chemotherapy) were observed for a maximum of 2.25 years in this study.
Arm/Group | Adjuvant or Metastatic Chemotherapy
Number analyzed (Participants) | 1121
Participants
  Profile 1 | 475
  Profile 2 | 439
  Profile 3 | 207

ADVERSE EVENTS:
Time Frame: Inclusion visit (Week 1) up to end of study visit (up to Week 19)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis was performed on safety population.
Arm/Group | Adjuvant Chemotherapy | Metastatic Chemotherapy
All-Cause Mortality (participants affected / at risk) | 2/552 | 41/608
Serious Adverse Events (participants affected / at risk) | 3/552 | 2/608
Other Adverse Events (participants affected / at risk) | 78/552 | 67/608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Chemotherapy (N=552) | Metastatic Chemotherapy (N=608)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Chemotherapy (N=552) | Metastatic Chemotherapy (N=608)
Nausea (Gastrointestinal disorders) | 11 | 10
Vomiting (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Anorexia (Gastrointestinal disorders) | 1 | 3
Mucite (Gastrointestinal disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
General physical health deterioration (General disorders) | 13 | 6
Injection site pain (General disorders) | 2 | 0
Allergic reaction (General disorders) | 1 | 0
Chest pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 44 | 29
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 2
Gamma-glutamyltransferase increased (Hepatobiliary disorders) | 0 | 2
Urinary track disorder (Renal and urinary disorders) | 1 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Asthenia (General disorders) | 1 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.